CLINICAL TRIAL: NCT05235919
Title: Repetitive Transcranial Magnetic Stimulation to Promote Helpful Self-regulatory Behaviour in Children and Youth With Autism Spectrum Disorder
Brief Title: Treatment to Promote Self-regulation in Children With Autism Spectrum Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Centre for Addiction and Mental Health (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Deryk Beal, Clinician-Scientist, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASDSR01
Record Dates: First submitted 2022-01-10; First posted 2022-02-11 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder; Self-Regulation, Emotion
Keywords: transcranial magnetic stimulation; rTMS; MRI
MeSH Terms: conditions — Autism Spectrum Disorder; Emotional Regulation | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized sham-controlled rTMS trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and outcomes assessor will be blind to rTMS or sham condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- repetitive transcranial magnetic stimulation (rTMS) (Experimental): Participants will receive 15 rTMS sessions for 3 weeks.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Sham (Sham Comparator): Participants will receive 15 sessions of sham stimulation for 3 weeks.
  Interventions: Other: Sham stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — 30 minutes rTMS session 5 days/week for 3 weeks.
  Arms: repetitive transcranial magnetic stimulation (rTMS)
Other: Sham stimulation — 30 minutes sham stimulation 5 days/week for 3 weeks.
  Arms: Sham

SUMMARY:
This study will evaluate the feasibility of repetitive Transcranial Magnetic Stimulation (rTMS) in Autism Spectrum Disorder (ASD) with self-regulation impairment. Baseline and follow-up participant visits will include behavioral assessments of self-regulation and magnetic resonance imaging (MRI) to determine neurophysiological outcomes before and after rTMS treatment.

DETAILED DESCRIPTION:
Children and youth with Autism Spectrum Disorder (ASD) often present with co-morbid impairments in self-regulation (e.g., difficulty managing their emotions) resulting in unhelpful regulatory approaches such as disruptive compulsive, aggressive and self-injurious behaviour. There is an urgent need to establish novel, precise and effective interventions that promote self-regulation and reduce disruptive behaviours. This project will collect pilot data on the effects of repetitive TMS in reducing disruptive behaviours in youth with ASD, in order to inform the design of a follow-up full-scale clinical trial. Youth with ASD who experience clinically significant difficulties with self-regulation and disruptive behaviour will be recruited. Participants will be randomized to rTMS or sham rTMS for 3 weeks. The overall feasibility of the trial will be assessed. The effect of rTMS on the brain mechanisms of self-regulation and clinical improvement in disruptive behaviours will also be measured. Neurophysiological outcomes, including changes in regional brain network activity for inhibition of behaviour, will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Children with a diagnosis of autism spectrum disorder and self-regulation impairment or challenges
* Able to participate in rTMS

Exclusion Criteria:

* Children with autism spectrum disorder but no co-morbid self-regulation disorders.
* Children with contraindications to TMS (history of seizures, family history of seizures, metal implants)
* Co-existing neurological conditions (epilepsy, stroke, etc.)

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Weeks 1-18
  Recruitment rates of 4 participants/month are achieved with a ≥ 20% response rate
Attrition | Weeks 1-18
  Attrition rates of less than 10% (i.e., ≥90% of participants successfully complete assessments).
Adherence | Weeks 1-18
  90% of participants who complete assessment achieve the target intensity and dose (15 rTMS sessions)
Blinding success | Weeks 1-18
  Blinding of participants and their parents/caregivers and required study team members will be assessed using a Blinding Questionnaire indicating the perceived group membership (rTMS/sham)

SECONDARY OUTCOMES:
Clinical Measure of Self-regulation: Emotion Dysregulation Index Reactivity and Dysphoria | Weeks 1, 6, 18
  Change in total score on Reactivity (0-96) and Dysphoria (0-24) scales - greater scores indicates a worse outcome
Clinical Measure of Self-Regulation: The Response To Stress Questionnaire - Family Stress | Weeks 1, 6, 18
  Change in total score Response To Stress Questionnaire Family Stress Version (57-228, greater score indicates worse a outcome)
Clinical Measure of Self-regulation: Aberrant Behaviour Checklist - Irritability Subscale | Weeks 1, 6, 18
  Change in total score on Aberrant Behaviour Checklist - Irritability Subscale (15-60, greater score indicates a worse outcome)
Clinical Measure of Self-regulation: Emotional Regulation Checklist | Weeks 1, 6, 18
  change in total score on Emotional Regulation Checklist (24-96, low scores indicate worse outcomes)
Overall Clinical Change | Weeks 1, 6, 18
  Clinical Global Impression scale - 1 item on a scale from 0-7 (a change of 0.5 indicates a clinical impact of significance)
Inhibitory control | Weeks 1, 6, 18
  Go/No-Go Task Performance
Functional brain changes (magnetic resonance imaging) | Weeks 1, 6, 18
  change in blood oxygen level dependent (BOLD) signal associated with go/no-go task
Structural brain changes (magnetic resonance imaging) | Weeks 1, 6, 18
  Diffusion imaging - change in fractional anisotropy

CONTACTS AND LOCATIONS:
Overall Officials: Deryk Beal, PhD, Principal Investigator — Holland Bloorview Research Institute
Locations (1):
- Bloorivew Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oberman LM, Enticott PG, Casanova MF, Rotenberg A, Pascual-Leone A, McCracken JT; TMS in ASD Consensus Group. Transcranial magnetic stimulation in autism spectrum disorder: Challenges, promise, and roadmap for future research. Autism Res. 2016 Feb;9(2):184-203. doi: 10.1002/aur.1567. Epub 2015 Nov 4. PMID 26536383